CLINICAL TRIAL: NCT00992758
Title: Phase I, Dose-Escalation Study of Iodine-131 Anti-B1 Antibody for Patients With Previously Treated Non Hodgkin's Lymphoma With More Than 25% Bone Marrow Involvement
Brief Title: Safety and Efficacy of Iodine-131 Anti-B1 Antibody for Non Hodgkin's Lymphoma (NHL) Patients With Greater Than 25% Bone Marrow Involvement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104512
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: bone marrow; Radioimmunotherapy; non-Hodgkin's lymphoma; Bexxar; anti-B1 antibody; tositumomab and iodine I-131 tositumomab; NHL; tositumomab
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tositumomab I-131

ARMS (1):
- Treatment, Non-Randomized, Open Label (Experimental): Treatment, Non-Randomized, Open Label, Uncontrolled, Single Group Assignment, Safety/Efficacy Study
  Interventions: Biological: Iodine-131 Anti-B1 Antibody

INTERVENTIONS:
Biological: Iodine-131 Anti-B1 Antibody — Dosimetric Dose: 450 mg unlabeled Anti-B1 Antibody infused over 1 hour or longer followed by 35 mg of Anti-B1 Antibody of which 1-2 mg has been labeled with 5 mCi of Iodine-131 infused over 20 minutes.
  Therapeutic Dose: 7-14 days after dosimetric dose, 450 mg Anti-B1 Antibody infused over 1 hour or longer followed by 35 mg of Anti-B1 Antibody labeled with the subject-specific dose of Iodine-131 to deliver the desired total body radiation, infused over 20 minutes The dose escalation will be initiated at 45 cGy and will be increased in 10 cGy increments until the maximum tolerated dose (MTD) is reached.
  Other Names: BEXXAR

SUMMARY:
This is a phase I, dose escalation, open-label, multicenter study of iodine-131 Anti-B1 Antibody for patients with non-Hodgkin's lymphoma (NHL) who have more than 25% bone marrow involvement with NHL. Prior studies with Iodine-131 Anti B1 Antibody for the treatment of NHL have excluded patients with more than 25% bone marrow involvement with NHL. To be eligible, patients must have been previously treated and failed to achieve an objective response on or relapse during or following their last treatment.

Patients will undergo two dosing phases while on study. In the first phase, termed the "dosimetric dose", patients will receive 450 mg unlabeled Anti-B1 Antibody infused over 1 hour or longer followed by 35 mg of Anti-B1 Antibody of which 1-2 mg has been labeled with 5 mCi of Iodine-131 infused over 20 minutes. Whole body camera scans will be obtained on Day 0, Day 2, 3, or 4, and Day 6 or 7 following the dosimetric dose. Using dosimetric data from three imaging time points, a patient-specific dose of Iodine-131 Anti-B1 Antibody to deliver the desired total body dose of radiotherapy will be calculated. In the second phase, termed the "therapeutic dose", 450 mg Anti-B1 Antibody will be infused over 1 hour or longer followed by 35 mg of Anti-B1 Antibody labeled with the subject-specific dose of Iodine-131 to deliver the desired total body radiation, infused over 20 minutes. The dose escalation will be initiated at 45 cGy and will be increased in 10 cGy increments until the maximum tolerated dose (MTD) is reached.

Patients will be treated with either saturated potassium iodide, Lugol's solution, or potassium iodide tablets starting at least 24 hours prior to the infusion of the dosimetric dose and continuing for 14 days following the last infusion of the therapeutic dose.

The primary endpoint is to determine the maximum tolerated dose of Iodine-131 Anti B-1 Antibody in patients with previously treated NHL having more than 25% bone marrow involvement with lymphoma. Secondary endpoints include assessment of response rate, duration of response, relapse-free survival, time to treatment failure, safety, and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed initial diagnosis of low-grade non-Hodgkin's B-cell lymphoma according to International Working Formulation (i.e., small lymphocytic [with or without plasmacytoid differentiation]; follicular small cleaved, or follicular, mixed small cleaved and large cell), or low-grade lymphoma that has transformed to a higher grade histology, or de novo follicular large cell lymphoma.
* Patients must have Ann Arbor Stage IV disease and greater than an average of 25% of the intratrabecular marrow space involved by NHL in bilateral bone marrow biopsy specimens as assessed microscopically at study entry. A unilateral bone marrow biopsy demonstrating greater than 50% involvement with NHL is also adequate for study entry.
* Patients must have been previously treated with chemotherapy and progressed on, failed to achieve an objective response on, or progressed after completion of their last chemotherapy.
* Patients must have evidence that their tumor tissue expresses the CD20 antigen.
* Patients must have a performance status of at least 60% on the Karnofsky Performance Scale and an anticipated survival of at least 3 months.
* Patients must have an ANC greater than 1500 cells/mm3 and a platelet count greater than or equal to 150,000 cells/mm3 within 14 days of study entry. These blood counts must be sustained without support of hematopoietic cytokines or transfusion of blood products.
* Patients must have adequate renal function (defined as serum creatinine less than 1.5 times the upper limit of normal) and hepatic function (defined as total bilirubin less than 1.5 times the upper limit of normal and AST less than 5 times the upper limit of normal) within 14 days of study entry.
* Patients must have bi-dimensionally measurable disease. At least one lesion must be greater than or equal to 2 x 2 cm.

Exclusion Criteria:

* Patients with active obstructive hydronephrosis.
* Patients with New York Heart Association class III or IV heart disease or other serious illness that would preclude evaluation.
* Patients with prior malignancy other than lymphoma, except for adequately treated skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 years. Patients who have been disease-free of another cancer for greater than 5 years must be carefully assessed at the time of study entry to rule out recurrent disease.
* Patients with known HIV infection.
* Patients who are HAMA positive.
* Patients with known brain or leptomeningeal metastases.
* Patients who have undergone therapy with either stem cell or bone marrow transplant.
* Patients who have received cytotoxic chemotherapy, immunosuppressants, or cytokine therapy within 4 weeks prior to study entry (6 weeks for nitrosourea compounds). The use of systemic steroids must be discontinued at least 1 week prior to study entry.
* Patients who are pregnant or breastfeeding. Patients of childbearing potential must undergo a serum pregnancy test within 7 days prior to study entry. Males and females must agree to use effective contraception for 6 months following the radioimmunotherapy dose.
* Patients with progressive disease within 1 year of irradiation arising in a field that has been previously irradiated with more than 3500 cGy.
* Patients who are concurrently receiving either approved or non-approved (through another protocol) anti-cancer drugs or biologics.
* Patients with active infection requiring IV anti-infectives at the time of study entry.
* Patients who have previously received radioimmunotherapy.
* Patients with de novo intermediate- or high-grade NHL, except for intermediate subtype of follicular large cell NHL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1999-05-28 (Actual); Primary Completion 2012-06-07 (Actual); Study Completion 2012-06-07 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of Iodine-131 Anti B-1 Antibody in patients with previously treated NHL having more than 25% bone marrow involvement with lymphoma. | Approximately 2 years

SECONDARY OUTCOMES:
response rate | Long term follow-up every 6 months
duration of response | Long term follow-up every 6 months
relapse-free survival | Long term follow-up every 6 months
time to treatment failure | Long term follow-up every 6 months
Safety as measured by adverse events, severity of hematologic toxicity, the use of supportive care and the percentage of human anti-murine antibody positivity | Long term follow-up every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 104512 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/104512?search=study&search_terms=104512#rs
- Available data/document: Individual Participant Data Set: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104512 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register